CLINICAL TRIAL: NCT04930432
Title: A Phase I/II Study of MCLA-129, a Human Anti-EGFR and Anti-c-Met Bispecific Antibody, in Patients With Advanced NSCLC and Other Solid Tumors, Evaluating Safety, Pharmacokinetic Characteristics and Antitumor Activity
Brief Title: Study of MCLA-129, a Human Bispecific EGFR and cMet Antibody, in Patients With Advanced NSCLC and Other Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTP-21711
Record Dates: First submitted 2021-05-31; First posted 2021-06-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumor; Non-Small Cell Lung Cancer; Head and Neck Cancer; Colorectal Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: dose escalation and dose expansion (Experimental): Participants will receive intravenous infusion of MCLA-129 every two weeks (Q2W) or every weeks (QW) at different dose in each dose level.
  Interventions: Drug: MCLA-129
- Part 2: cohort expansion (Experimental): Participants will receive intravenous infusion of MCLA-129 every two weeks (Q2W) at the recommended Phase II dose (RP2D) in each cohort.
  Interventions: Drug: MCLA-129

INTERVENTIONS:
Drug: MCLA-129 — MCLA-129 will be administered by intravenous infusion on the 28-day treatment cycle.

SUMMARY:
This is a multi-center, open-label, Phase I/II clinical study of MCLA-129 as monotherapy in patients with advanced solid tumors to evaluate the safety, pharmacokinetic characteristics and antitumor activity of MCLA-129.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-agent phase I/II clinical study of MCLA-129 in patients with advanced solid tumors to evaluate the safety, pharmacokinetic profile, and antitumor activity of MCLA-129. The study consists of two parts: Part I is a phase I dose- finding study in patients with advanced solid tumors, including a dose escalation phase and a dose expansion phase; Part II is a phase II parallel cohort expansion study to further evaluate the efficacy, safety and PK profile of MCLA-129 in sub-cohorts of patients with advanced non-small cell lung cancer and other solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are ≥ 18 years of age, regardless of gender.
* Subjects must have histologically or cytologically confirmed metastatic or unresectable advanced NSCLC or other solid tumors (including but not limited to head and neck cancer, colorectal cancer, etc.), have disease progression after standard treatment, or are intolerant to standard treatment, or refuse standard treatment (Refusal of standard treatment does not apply to Part 2).
* For Part 1, subjects must be diagnosed with EGFR positive and/or MET positive by testing.

For patients with advanced NSCLC, EGFR positive is defined as: EGFR mutation or EGFR amplification. MET positive is defined as: MET amplification or MET exon 14 skipping mutation.

For patients with other advanced solid tumors other than NSCLC, EGFR positive is defined as: High EGFR expression or EGFR amplification. MET positive is defined as: c-Met high expression or MET amplification.

• For Part 2, patients shall meet the inclusion criteria for each cohort by biomarker testing.

Cohort A: Patients with advanced NSCLC who are previously diagnosed with EGFR mutations and treated with third-generation EGFR-TKIs for drug resistance.

Cohort B: Advanced NSCLC patients diagnosed with EGFR exon 20 insertion mutation (Exon20ins).

Cohort C: Advanced NSCLC patients with MET amplification. Cohort D: Advanced NSCLC patients with MET exon 14 skipping mutation (Exon14 skipping).

Cohort E: Patients with locally advanced or recurrent metastatic colorectal cancer (CRC) could not undergo curative treatment.

Cohort F: Other advanced solid tumors that have failed or are intolerant to standard therapy.

Cohort G: Patients with locally advanced or metastatic MET-amplified or MET-overexpressing other driver gene-negative non-small cell lung cancer, gastric/gastroesophageal junction adenocarcinoma [including signet ring cell carcinoma, mucinous adenocarcinoma, and hepatoid adenocarcinoma], or recurrent/metastatic [R/M] head and neck squamous cell carcinoma [primary sites: oral cavity, oropharynx, hypopharynx, or larynx], who are not candidates for curative treatment.

* For subjects in the dose escalation phase of Part 1, evaluable lesions must be present; other subjects must have measurable lesions that meet the definition of RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Expected survival ≥3 months.
* Have adequate organ function (no blood transfusion or use of blood component or G-CSF support within 14 days before testing).
* Willing and able to follow the trial and follow-up procedures.
* Able to understand the nature of the trial and voluntarily sign the written informed consent form.

Exclusion Criteria:

* For colorectal cancer subjects, HER-2 positivity (IHC 2+/3+ or FISH/NGS+) confirmed by local or central laboratory genetic testing.
* Have received an investigational product or anti-tumor drug treatment within 14 days before the first dose of MCLA-129 or within 5 half-lives of the drug (whichever is longer). For cohort E1, the interval between the last dose of EGFR monoclonal antibody and the first dose of MCLA-129 was less than 6 months.
* Have undergone a major surgery and radiotherapy (local palliative radiotherapy is allowed 2 weeks or more prior to the first dose) within 4 weeks prior to the first dose of MCLA-129.
* For patients with colorectal cancerr, head and neck squamous cell carcinoma, or gastric/gastroesophageal junction adenocarcinoma: patients who have previously received systemic anti-tumor therapy beyond the third line (excluding maintenance therapy).
* For subjects with non-small cell lung cancer only: have received more than 2 prior lines of cytotoxic chemotherapy for locally advanced or metastatic diseases (excluding maintenance therapy).
* For advanced NSCLC patients with EGFR Exon20ins mutation: have received prior EGFR-TKI therapy (e.g., poziotinib, TAK-788, DZD9008, CLN-081, or furmonertinib, etc.) that is known to be effective against Exon20ins.
* Prior use of EGFR/c-Met bispecific antibody or ADC drugs (such as Amivantamab, EMB-01, GB263T, PM1080/HS-20117, TAVO412, YH013/ DM005, SHR-9839 or AZD9592 etc.).
* Prior to the first dose of MCLA-129, previous treatment-related toxicities have not resolve to Grade 1 or below (CTCAE 5.0 criteria), except for alopecia.
* Have had other malignancies within the past 3 years, except for cancers that have been totally cured or locally cured, such as basal or squamous cell carcinoma of the skin, cervical cancer in situ, or breast cancer in situ.
* Patients with primary malignant tumor of central nervous system, or metastases to meninges, spinal cord compression, or at risk of cerebral hemorrhage, or concomitantly with symptomatic brain metastases, or new therapy naive brain metastases. For cohorts E, F and G (excluding NSCLC patients): Patients with known brain metastases and/or meningeal metastases, or primary malignant tumor of central nervous system. Subjects with neurological symptoms shall have a brain CT/MRI scan to exclude brain metastases.
* With clinically significant cardiovascular and cerebrovascular diseases.
* Active hepatitis B (positive hepatitis B surface antigen (HBsAg) or core antibody (HBcAb) and serum HBV DNA ≥ 2,000 IU/mL [equivalent to 104 copies/mL]), positive hepatitis C virus antibody, HIV antibody and treponema pallidum antibody.
* Subjects with a history of interstitial lung disease or current clinical evidence of interstitial lung disease, including drug-induced Interstitial lung disease, radiation pneumonitis or pulmonary fibrosis. Subjects who could not be ruled out for suspected interstitial lung disease/pulmonary fibrosis through imaging examinations during screening, or those with uncontrolled/unstable non-infectious pneumonitis/pulmonary inflammation are excluded.
* Presence of a serious disease or medical condition currently, including but not limited to uncontrolled active infection, uncontrolled pleural or peritoneal effusion, unstable/uncontrolled tuberculosis, active gastrointestinal diseases, gastrointestinal obstruction or perforation risks, and clinically significant pulmonary, metabolic or psychiatric diseases.
* Females of childbearing potential, pregnant or breastfeeding women with a positive serum pregnancy test 7 days before the start of treatment, and male and female subjects who are unwilling to use effective contraceptive measures or plan to have a child throughout the treatment period and within 3 months after the end of treatment.
* Patients with known allergic reactions and hypersensitivity reactions, or be allergic to MCLA-129 or any of its excipients.
* Patients with poor compliance, inability or unwillingness to follow the study and/or follow-up procedure listed in the protocol, or patients who are not suitable to participate in this trial, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) in Part 1 | First 28 days of treatment
  To determine the dose-limiting toxicity (DLT) of single agent MCLA-129 in patients with advanced solid tumors in Part 1.
Maximum Tolerated Dose (MTD) in Part 1 | First 28 days of treatment
  To determine the maximum tolerated dose (MTD) of single agent MCLA-129 in patients with advanced solid tumors in Part 1.
Overall Response Rate (ORR) in Part 2 | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years
  To evaluate the efficacy of MCLA-129 at RP2D in patients with advanced NSCLC and other solid tumors in each cohort in Part 2 in terms of overall response rate (ORR)
Treatment-Emergent Adverse Event (TEAE) in Part 1 and 2 | Until 30 days after the last dosing
  To evaluate the safety of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of treatment-emergent adverse event (TEAE)

SECONDARY OUTCOMES:
Half-life [t1/2] in Part 1 and 2 | Until 30 days after the last dosing
  To evaluate the population PK profile of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of half-life (t1/2)
Apparent volume of distribution [VSS] in Part 1 and 2 | Until 30 days after the last dosing
  To evaluate the population PK profile of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of apparent volume of distribution [VSS]
Maximum plasma concentration [Cmax] in Part 1 and 2 | Until 30 days after the last dosing
  To evaluate the population PK profile of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of maximum plasma concentration [Cmax]
Time to reach maximum concentration [Tmax] in Part 1 and 2 | Until 30 days after the last dosing
  To evaluate the population PK profile of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of time to reach maximum concentration [Tmax]
Area under the concentration versus time curve from time zero to time t [AUC0-t] in Part 1 and 2 | Until 30 days after the last dosing
  To evaluate the population PK profile of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of area under the concentration versus time curve from time zero to time t [AUC0-t]
Area under the concentration versus time curve [AUC0-∞] in Part 1 and 2 | Until 30 days after the last dosing
  To evaluate the population PK profile of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of area under the concentration versus time curve [AUC0-∞]
Overall Response Rate (ORR) in Part 1 | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years
  To evaluate the efficacy of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 in terms of overall response rate (ORR)
Disease Control Rate (DCR) in Part 1 and 2 | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years
  To evaluate the efficacy of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of disease control rate (DCR)
Progression-Free Survival (PFS) in Part 1 and 2 | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years
  To evaluate the efficacy of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of progression-free survival (PFS)
Clinical benefit rate (CBR) in Part 1 and 2 | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years
  To evaluate the efficacy of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of clinical benefit rate (CBR)
Duration of Response (DOR) in Part 1 and 2 | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years
  To evaluate the efficacy of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of duration of response (DOR)
Time to response (TTR) in Part 1 and 2 | From date of first treatment every 6 weeks until disease progression, death or withdrawal, whichever came first, approximately 2 years
  To evaluate the efficacy of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of time to response (TTR)
Overall Survival (OS) in Part 1 and 2 | From date of first treatment every 6 weeks until death or withdrawal, whichever came first, approximately 2 years
  To evaluate the efficacy of MCLA-129 in patients with advanced NSCLC and other solid tumors in Part 1 and 2 in terms of overall survival (OS)
Anti-Drug Antibody (ADA) in Part 1 and 2 | Until 30 days after the last dosing
  To assess the Incidence of anti-drug antibodies in serum blood against MCLA-129 following administration of MCLA-129
Cytokines in Part 1 | Before and after each administration on day 1 and day 15
  To assess the changes in cytokine levels in serum blood following administration of MCLA-129

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, PhD, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (87):
- China (87):
  - Affiliated Hospital of Hebei University, Baoding
  - Beijing Cancer Hospital, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Beijing Tongren Hospital, Beijing
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking University International Hospital, Beijing
  - The Fifth Medical Center of PLA Ceneral Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu
  - Cangzhou Hospital of Integrated TCM-WM·Hebei, Cangzhou
  - Ji Lin Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - The Second Xiangya Hospital of Central South University, Changsha
  - Xiangya Hospital of Central South University, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - Chifeng Municipal Hospital, Chifeng
  - Army Medical Center of PLA, Chongqing
  - Chongqing University Cancer Hospital, Chongqing
  - China-Japan Union Hospitai Of Jilin University, Ch’ang-ch’un
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - Fujian Cancer Hospital, Fuzhou
  - Fuzhou Pulmonary Hospital of Fujian, Fuzhou
  - The 900 Hospital of the Joint Service Support Force of the People's Liberation Army of China, Fuzhou
  - First Affiliated Hospital Of Gannan Medical University, Ganzhou
  - Guangdong Province Traditional Chinese Medical Hospital, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - The Frist Affiliated Hospital of Guangzhou Medical College, Guangzhou
  - The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Cancer Hospital of The University of Chinese Academy of Sciences, Hangzhou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Hanzhong Central Hospital, Hanzhong
  - Harbin Medical University Cancer Hospital, Harbin
  - Cancer Hospital affiliated to Harbin Medical University, Ha’erbin
  - Harbin Medical University cancer hospital, Ha’erbin
  - The Second Hospital of Anhui Medical University, Hefei
  - Henan Cancer Hospital (Affiliated Cancer Hospital of Zhengzhou University), Henan
  - Inner Mongolia People's Hospital, Hohhot
  - Jiangxi cancer hospital, Jiangxi
  - The First Hospital of Jilin University, Jilin
  - Shandong Cancer Hospital & institute, Jinan
  - Yunnan Cancer Hospital, Kunming
  - The First Hospital of Lanzhou University, Lanzhou
  - Jiangxi Cancer Hospital, Nanchang
  - General Hospital of Eastern Theater Command, Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - Nanjing Drum Tower Hospital, Nanjing
  - Guangxi Medical University Cancer Center, Nanning
  - Nantong Tumor Hospital, Nantong
  - Qingdao Central Hospital, Qingdao
  - The Affiliated Hospital of Qingdao University, Qingdao
  - First Hospital of Qinhuangdao, Qinhuangdao
  - ShangHai Chest Hospital, Shanghai
  - Shanghai Ninth People's Hospital, Shanghai JiaoTong University School of Medicine, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - Liaoning Cancer Hospital & Institute, Shenyang
  - Liaoning Cancer Hospital, Shenyang
  - The First Hospital of China Medical University, Shenyang
  - Cancer Hospital of Chinese Academy of Medical Sciences Shenzhen Hospital, Shenzhen
  - Shenzhen People's Hospital, Shenzhen
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Shanxi Provincial Cancer Hospital, Taiyuan
  - Taizhou Hospital of Zhejiang Province, Taizhou
  - General Hospital of Tianjin Medical University, Tianjin
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Tonghua Central Hospital, Tonghua
  - Weifang People's Hospital, Weifang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Hubei Cancer Hospital, Wuhan
  - Renmin Hospital of Wuhan University/Hubei General Hospital, Wuhan
  - Union Hospital, Tongji Medical College Huazhong University of Science and Technolog, Wuhan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Zhongnan Hospital Affiliated to Wuhan University, Wuhan
  - The First Affiliated Hospital of Wannan Medical College (Yijishan Hospital), Wuhu
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital Of Xiamen University, Xiamen
  - Xuzhou Central Hospital, Xuzhou
  - Yantai Yuhuangding Hospital, Yantai
  - The No. 2 People's Hospital of Yibin Sichuan, Yibin
  - Hospital of Ningxia Medical University, Yinchuan
  - He Nan Cancer Hospital, Zhengzhou
  - Henan Provincial People's Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Henan Provincial People's Hospital, Zhenzhou

IPD SHARING:
Plan to Share IPD: No